CLINICAL TRIAL: NCT06082258
Title: Evaluation of a Training and Support Intervention for General Practitioners Managing Patients With Persistent Symptoms Following a COVID-19 Episode
Brief Title: Education of Medical Staff to Post Acute Covid susTained sYmptoms
Acronym: EMPATY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Health Services Research
Other Study IDs: APHP220136; ECTZ199383 (Other Grant/Funding Number: ANRS/MIE); 2022-A00531-42 (Registry Identifier: IDRCB); DR-2023-132 (Other: Commission Nationale de l'Informatique et des Libertés)
Record Dates: First submitted 2023-10-12; First posted 2023-10-13 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Post-acute COVID-19 Syndrome
Keywords: Long COVID; Post acute Covid syndrome; Somatic symptom disorder; Education
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- usual care (No Intervention): Patients followed by general practitioners with no specific education on long COVID or somatic symptom disorders
- intervention (Experimental): Patients followed by general practitioners who have received a training in long COVID and somatic symptom disorders diagnosis and treatment, with reimbursement of three long consultations
  Interventions: Other: Training in the management of functional disorders; Other: Reimbursement of 3 long consultations

INTERVENTIONS:
Other: Training in the management of functional disorders — Theoritical and practical training of GP in long COVID and somatic symptom disorders management
  Arms: intervention
Other: Reimbursement of 3 long consultations — 3 long consultations (1 hour) reimbursed for each patient
  Arms: intervention

SUMMARY:
Evaluation of the effectiveness of a training and support intervention for general practitioners treating patients with persistent symptoms after a COVID-19 episode on the patients'quality of life at 3 months.

DETAILED DESCRIPTION:
Apart from the objectivable sequelae of a severe COVID-19 episode, the pathophysiology of symptoms persisting several months after an acute COVID episode is not established. The investigators hypothesize that a substantial part of these symptoms are functional somatic disorders, defined by symptoms not explained by a lesion of the organ which they designate and which can benefit from an action on their cognitive and behavioural mechanisms including an adapted physical activity program. The frequency of these symptoms and their major impact justifies the development of an adapted care offer easily accessible, involving mainly general practitioners (GP). For example, the ARS has advocated for the development of "covid-long" support cells, whose role is to coordinate the management of patients with these symptoms by providing advice and referral to other professionals if necessary. Experience has shown that doctors are baffled by the very polymorphic symptomatology of these patients and often have difficulty managing their anxiety towards the symptoms.

Primary Objective:

Describe the impact of GP training accompanied by a Covid Long Support Cell (CACL) to manage persistent somatic functional symptoms attributed to COVID-19 on the quality of life of patients at 3 months.

The main criterion of evaluation will be the evolution of the SF-12 quality of life physical composite score at 3 months.

Methods:

Prospective observational study. An observation phase before training during which the monitoring of 4 to 6 patients by general practitioners will be carried out according to the usual care management. Subsequently, general practitioners will be trained (intervention) and after training, 4 to 6 patients per general practitioner will then be recruited. The intervention will include:

1. Training delivered to CACL staff and volunteer general practitioners: online theoretical courses and video capsules produced with actors, discussed with learners, an expert doctor and an expert patient (several training sessions will be organized during the study).
2. Reimbursement for each patient of 3 long consultations (1 hour) with a participating general practitioner and an assessment by an adapted physical activity teacher during the first month of the patient's participation.
3. Follow-up of the patient by telephone interview at inclusion then at 1, 3 and 6 months after inclusion: physical and mental components of the SF-12, intensity of symptoms; healthcare consumption, work stoppage, physician satisfaction and patient experience, 1, 3 and 6 months.

Study population: patients managed by one of the 6 CACL of Ile de France.

Statistical Analysis:

The objective of the study is to describe the impact of the training of private general practitioners, accompanied by a support and coordination unit, for the management of persistent functional somatic symptoms attributed to COVID-19, on the quality of life linked to the physical health of patients at 3 months. The number of subjects to be included is set at 400 to be able to examine the results with sufficient precision within an acceptable time frame taking into account the expected rate of inclusion of approximately 1 patient per month, per general practitioner over a period of 14 months.

Assuming an average SF-12 SCP at 3 months of 31 in the control group with a standard deviation of 8 based on the results of the SF-12 questionnaire carried out in a sample of 216 patients with long COVID having consulted at the Hôtel-Dieu, a total of 400 patients will demonstrate an average SF-12 SCP at 3 months of 34 in the experimental group, with an alfa risk of 5% and a power of 96%.

The study will be systematically offered to all patients referred by their treating physician or who refer themselves to a CACL for prolonged symptoms attributed to "long COVID", this will best ensure good representativeness of the sample.

The SCP of the SF-12 questionnaire at 3 months will be compared between the patients included before and after the training using a mixed linear regression, taking into account in the model a random effect on the general practitioner and the adjustment on the SCP at inclusion.

The secondary objectives will also be analyzed using appropriate mixed models depending on the type of variables analyzed, considering the general practitioner as a random effect.

ELIGIBILITY:
Inclusion Criteria:

* at least two symptoms attributed to COVID-19 (including fatigue, dyspnea, cognitive impairment or pain); persistent for more than 2 months; not explained by a diagnosis unrelated to COVID-19;
* a quality of life impairment considered significant by the patient.

Exclusion Criteria:

* Refusal to participate in the study
* Under 18 years of age
* Persistent symptoms secondary to an objective sequelae from the initial episode of COVID-19.
* Neuropsychiatric disorder that may impair cognitive function prior to COVID-19
* Medical contraindication to physical training (pericarditis or myocarditis...)
* Patient not affiliated with the social security system or under AME
* Patient under guardianship, guardianship or guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change of physical component summary (PCS) of 12-Item Short-Form Health Survey (SF-12v2) - quality of life scale at 3 months compared to the PCS at the inclusion of the patient | 3 months
  Health-related quality of life variable measured using the Short Form Health Survey (SF-12v2): 12-item self-report that assesses physical and mental health related quality of life. The physical component summary (PCS) will be used. Normalized score ranges from 0 to 100, with higher scores indicating better physical health functioning.

SECONDARY OUTCOMES:
Change of physical component summary (PCS) of 12-Item Short-Form Health Survey (SF-12v2) - quality of life scale at 1 month compared to the PCS at the inclusion of the patient | 1 month
  Health-related quality of life variable measured using the Short Form Health Survey (SF-12v2): 12-item self-report that assesses physical and mental health related quality of life. The physical component summary (PCS) will be used. Normalized score ranges from 0 to 100, with higher scores indicating better physical health functioning.
Change of physical component summary (PCS) of 12-Item Short-Form Health Survey (SF-12v2) - quality of life scale at 6 months compared to the PCS at the inclusion of the patient | 6 months
  Health-related quality of life variable measured using the Short Form Health Survey (SF-12v2): 12-item self-report that assesses physical and mental health related quality of life. The physical component summary (PCS) will be used. Normalized score ranges from 0 to 100, with higher scores indicating better physical health functioning.
Change of mental component summary (MCS) of 12-Item Short-Form Health Survey (SF-12v2) - quality of life scale at 1 month compared to the MCS at the inclusion of the patient | 1 month
  Health-related quality of life variable measured using the Short Form Health Survey (SF-12v2): 12-item self-report that assesses physical and mental health related quality of life. The mental component summary (MCS) will be used. Normalized score ranges from 0 to 100, with higher scores indicating better mental health functioning.
Change of mental component summary (MCS) of 12-Item Short-Form Health Survey (SF-12v2) - quality of life scale at 3 months compared to the MCS at the inclusion of the patient | 3 months
  Health-related quality of life variable measured using the Short Form Health Survey (SF-12v2): 12-item self-report that assesses physical and mental health related quality of life. The mental component summary (MCS) will be used. Normalized score ranges from 0 to 100, with higher scores indicating better mental health functioning.
Change of mental component summary (MCS) of 12-Item Short-Form Health Survey (SF-12v2) - quality of life scale at 6 months compared to the MCS at the inclusion of the patient | 6 months
  Health-related quality of life variable measured using the Short Form Health Survey (SF-12v2): 12-item self-report that assesses physical and mental health related quality of life. The mental component summary (MCS) will be used. Normalized score ranges from 0 to 100, with higher scores indicating better mental health functioning.
Change of clinical global impression (CGI scores) of the patient at 1 month compared to the last available clinical evaluation | 1 month
  The CGI questionnaire is rated on a 7-point scale and score ranges range from 1 (very much improved) through to 7 (very much worse). Each component of the CGI is rated separately.
  The following components will be considered: fatigue, pain, breathing difficulties, attention and concentration problems, other persistent symptoms.
Change of clinical global impression (CGI scores) of the patient at 3 months compared to the last available clinical evaluation | 3 months
  The CGI questionnaire is rated on a 7-point scale and score ranges range from 1 (very much improved) through to 7 (very much worse). Each component of the CGI is rated separately.
  The following components will be considered: fatigue, pain, breathing difficulties, attention and concentration problems, other persistent symptoms.
Change of clinical global impression (CGI scores) of the patient at 6 months compared to the last available clinical evaluation | 6 months
  The CGI questionnaire is rated on a 7-point scale and score ranges range from 1 (very much improved) through to 7 (very much worse). Each component of the CGI is rated separately.
  The following components will be considered: fatigue, pain, breathing difficulties, attention and concentration problems, other persistent symptoms.
Frequency of patient care consultations at 1 month | 1 month
  Number of patient care consultations between inclusion and 1-month follow-up
Frequency of patient care consultations at 3 months | 3 months
  Number of patient care consultations between inclusion and 3-month follow-up
Frequency of patient care consultations at 6 months | 6 months
  Number of patient care consultations between inclusion and 6-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte Ranque, Pr, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (7):
- France (7):
  - Paris Nord (CPTS 10e), Paris
  - Paris Est (CPTS 12e et 20e), Paris
  - DAC 75, Paris
  - Paris Sud (CPTS 13-14e), Paris
  - Paris Ouest (CPTS 15e), Paris
  - DAC 93, Saint-Denis
  - DAC 92, Suresnes

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in publication could be shared. IPD detailed in the protocol of a planned metaanalysis could be shared
Supporting Information: Study Protocol, ICF
Time Frame: Two years after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on a scientific project and scientific involvement of the PI team. Collaboration will be fostered. Data sharing must respect the agreements made with funders. Teams wishing obtain IPD must meet the sponsor and IP team to present scientific (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractual agreement.
  Processing of shared data must comply with European General Data Protection Regulation (GDPR).